CLINICAL TRIAL: NCT06936709
Title: Effect of Colchicine in the Perioperative Period on Reducing Post-Operative Pain in Total Knee Arthroplasty
Brief Title: Perioperative Colchicine for TKA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: St. Luke's Hospital, Kansas City, Missouri (Other)
Responsible Party: Principal Investigator, John Mercuri, MD, Medical Doctor, Geisinger Clinic
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-0488
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis of Knee; Recovery Following Primary Total Knee Arthroplasty; Perioperative Pain Control
Keywords: Total Knee Arthroplasty; Colchicine; Postoperative Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Colchicine Loading Dose Only (Experimental): Patients in this arm will receive 1.8 mg of colchicine on postoperative day 0. This dosage aligns with standard of care loading dose for acute gout attacks. This will be a one time dosage of colchicine. On postoperative days 1-3, patients will take placebo dextrose pills twice daily.
  Interventions: Drug: Colchicine 1.8 mg (loading dose) + Dextrose Oral Placebo
- Colchicine Loading Dose + Maintenance Dose (Experimental): Patients in this arm will receive a 1.8 mg loading dose of colchicine on postoperative day 0. They will then take a 0.6 mg maintenance dose twice daily on postoperative days 1-3. This dosage of colchicine in this arm models standard of care dosing for acute gout attacks.
  Interventions: Drug: Colchicine 1.8 mg + 0.6 mg
- Placebo Group (Placebo Comparator): Patients in this arm will receive a placebo dextrose pill on postoperative day 0. They will then take a placebo dextrose pill twice daily on postoperative days 1-3.
  Interventions: Drug: Dextrose Oral Placebo

INTERVENTIONS:
Drug: Colchicine 1.8 mg (loading dose) + Dextrose Oral Placebo — This intervention will be used for individuals in arm A of the study who will receive a loading dose of colchicine (1.8 mg) on postoperative day 0, and will then be given placebo oral dextrose pills to take twice daily on postoperative days 1-3
  Arms: Colchicine Loading Dose Only
Drug: Colchicine 1.8 mg + 0.6 mg — This intervention is will be given to patients in arm B of the study who will receive a loading dose of colchicine (1.8 mg) on postoperative day 0, followed by a maintenance does of colchicine (0.6 mg) to be taken twice daily on postoperative days 1-3.
  Arms: Colchicine Loading Dose + Maintenance Dose
Drug: Dextrose Oral Placebo — This intervention will be for patients in arm C, the placebo arm. These patients will receive oral dextrose pills to be taken once on postoperative day 0, and twice daily on postoperative days 1-3.
  Arms: Placebo Group

SUMMARY:
This study is a prospective, randomized, double-blinded, placebo-controlled study of the drug colchicine in the acute postoperative period for patients who are undergoing a total knee arthroplasty (TKA). Patients aged 18 years or older who are undergoing TKA will be invited to participate in the study. The primary endpoint of this study is to determine if colchicine, an anti-inflammatory medication commonly used for gout attacks, will decrease the postoperative pain of patients undergoing elective TKA.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blinded, placebo-controlled study of the drug colchicine in the acute postoperative period for patients who are undergoing a total knee arthroplasty (TKA). Patients aged 18 years or older who are undergoing TKA will be invited to participate in the study. The primary endpoint of this study is to determine if colchicine, an anti-inflammatory medication commonly used for gout attacks, will decrease the postoperative pain of patients undergoing TKA.

In doing so, we will utilize a 3-arm approach with two experimental groups and one placebo group. Qualifying subjects will be randomized 1:1:1 to Group A receiving a 1.8 mg loading dose of colchicine, Group B receiving the same loading dose + 0.6 mg maintenance dose of colchicine to be taken twice daily, and Group C receiving a placebo.

Regarding study procedures, standard preoperative and intraoperative procedures will be employed to ensure experimental and control groups have a nearly equivalent experience before the intervention. Subjects will be discharged with the same ambulation instructions and physical therapy regimens. Aside from the experimental drug, patients will receive the same postoperative pain medications upon discharge.

Research staff in the Geisinger pharmacy will receive and prepare the oral medication for dispensing, which will include randomizing identification numbers to colchicine or placebo, labeling packages with study identification numbers and subject information, and ensuring there is no visible method to discern colchicine from placebo. Colchicine is to be stored at room temperature.

Providers and subjects will be blinded regarding whether the subject will receive a colchicine loading dose + the placebo pills for maintenance doses, a colchicine loading dose + colchicine for maintenance doses, or the placebo pills for both. Group A will receive a 1.8 mg loading dose of colchicine by mouth on postoperative day 0 and will be instructed to take a placebo by mouth twice daily on postoperative days 1-3. Group B will receive a 1.8 mg loading dose of colchicine by mouth on postoperative 0 and will be instructed to take a 0.6 mg maintenance dose of colchicine by mouth twice daily on postoperative days 1-3. Group C will receive placebo dextrose pills by mouth on postoperative day 0 and will be instructed to take the placebo by mouth twice daily on postoperative days 1-3. Subjects will be sent home with an adequate supply of pills for postoperative days 1-3 and instructions on use.

The procedure for measuring the study variables is as follows:

Subjects will receive a post-operative pain journal upon hospital discharge on postoperative day 0. The journal will include three time points (morning, midday, and bedtime) in which they will record a VAS pain score ranging from 0-10 for post-operative days 1-3. The journal will also include a box for subjects to record the total pills of the prescribed postoperative opioid they have taken each day on postoperative days 1-3. Lastly, the journal will include a checkbox at the end for subjects to record whether they have experienced known colchicine-related side effects on postoperative days 1-3 such as nausea, vomiting, diarrhea, and abdominal pain. For evaluation of KOOS-JR scores and knee flexion, subjects will complete the 7-question KOOS-JR questionnaire at their 2-, 6-, and 12-week post-operative visits, and at these visits, a member of the research staff will determine the subject's knee flexion. Lastly, regarding the assessment of 90-day postoperative complications, the researchers will conduct a review of the subject's EHR.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older undergoing elective total knee arthroplasty for osteoarthritis.

Exclusion Criteria:

* Subject has impaired hepatic function (Child-Pugh Class >B)
* Subject has impaired renal function (GFR < 60 ml/min/1.73 m2)
* Subject has known adverse reaction to colchicine
* Subject has chronic opioid use (Filled opioid medication twice within 6 months of surgical date)
* Subject is pregnant or expecting to become pregnant during the time of the study associated with colchicine exposure (postoperative days 0-3)
* Subject is unable to provide informed consent
* Subject is actively prescribed medication that interact with colchicine in a manner that would increase the risk of colchicine toxicity, i.e.:
* Antifungals: Ketoconazole, itraconazole, fluconazole, etc…
* Macrolides : Clarithromycin, erythromycin
* HIV protease : Ritonavir, Atazanavir, saquinavir, etc...
* Ca2+: Verapamil and Diltiazem
* Cyclosporine
* Danazol
* Amiodorone
* Quinidine
* Anti-hepaciviral combinations
* Grapefruit juice
* Statins: atorvastatin, lovastatin, simvastatin, etc…
* Gemfibrozil and other fibrates
* Digoxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative VAS pain score | From postoperative day 0 through postoperative day 4.
  Subjects will receive a post-operative pain journal upon hospital discharge on postoperative day 0. The journal will include three time points (morning, midday, and bedtime) in which they will record a VAS pain score ranging from 0-10 for post-operative days 1-3. 0 being no pain, 10 being the worst pain they have ever experienced.

SECONDARY OUTCOMES:
Daily Opioid Usage | From postoperative day 0 through postoperative day 3.
  Subjects will receive a post-operative pain journal upon hospital discharge on postoperative day 0. The journal will include three time points (morning, midday, and bedtime) in which they will record the total pills of the prescribed postoperative opioid they have taken each day on postoperative days 1-3.
Postoperative KOOS-JR Score | From postoperative day 0 through postoperative week 12.
  Subjects will complete the 7-question KOOS-JR questionnaire at their 2-, 6-, and 12-week post-operative visits. Scoring ranges from 0-28, measuring variables from 0 (none) to 4 (extreme). Questions asked are: How severe is your knee stiffness after first wakening in the morning? What amount of knee pain have you experienced the last week during the following activities?
  * Twisting/pivoting on your knee
  * Straightening knee fully
  * Going up or down stairs
  * Standing upright And the what degree of difficulty have you had with the following activities?
  * Rising from sitting
  * Bending to floor/pick up an object
Postoperative Knee Flexion | Postoperative day 0 through postoperative week 12.
  Subject's knee flexion will be assessed at their 2-, 6-, and 12- week postoperative visits to assess recovery from their TKA. Values will be recording in degree of flexion, representing their range of motion.
90 day postoperative complications | Postoperative day 0 to postoperative day 90
  Subject's 90-day postoperative complications such as ED visits, unplanned readmission, joint infection, wound dehiscence, deep vein thrombosis, pulmonary embolism, or return to OR, etc. Assessment of these complications will be done through a chart review of the subject's electronic health records.
Colchicine Related Side Effects | Postoperative day 0 through postoperative day 3.
  The assessment of colchicine related side effects such as diarrhea, vomiting, abdominal pain, nausea, fatigue, headache, and pharyngolaryngeal pain will be recorded by subjects in the postoperative journal that they will receive on postoperative day 0. A checkbox will be present for each known side-effect for patients to self-report if they have had any of the aforementioned symptoms.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nazia, S, Robinson, K, Terrell, J. Colchicine. StatPearls Publishing. Updated January 2025. Accessed March 20, 2025., https://www.ncbi.nlm.nih.gov/books/NBK431102/
- [Background] Danoff JR, Goel R, Sutton R, Maltenfort MG, Austin MS. How Much Pain Is Significant? Defining the Minimal Clinically Important Difference for the Visual Analog Scale for Pain After Total Joint Arthroplasty. J Arthroplasty. 2018 Jul;33(7S):S71-S75.e2. doi: 10.1016/j.arth.2018.02.029. Epub 2018 Feb 22. PMID 29567002
- [Background] Huang ZY, Huang Q, Wang LY, Lei YT, Xu H, Shen B, Pei FX. Normal trajectory of Interleukin-6 and C-reactive protein in the perioperative period of total knee arthroplasty under an enhanced recovery after surgery scenario. BMC Musculoskelet Disord. 2020 Apr 21;21(1):264. doi: 10.1186/s12891-020-03283-5. PMID 32316949
- [Background] Heijman MWJ, Fiolet ATL, Mosterd A, Tijssen JGP, van den Bemt BJF, Schut A, Eikelboom JW, Thompson PL, van den Ende CHM, Nidorf SM, Popa CD, Cornel JH. Association of Low-Dose Colchicine With Incidence of Knee and Hip Replacements : Exploratory Analyses From a Randomized, Controlled, Double-Blind Trial. Ann Intern Med. 2023 Jun;176(6):737-742. doi: 10.7326/M23-0289. Epub 2023 May 30. PMID 37247416
- [Background] Shvartz V, Le T, Enginoev S, Sokolskaya M, Ispiryan A, Shvartz E, Nudel D, Araslanova N, Petrosyan A, Donakanyan S, Chernov I, Bockeria L, Golukhova E. Colchicine in Cardiac Surgery: The COCS Randomized Clinical Trial. J Cardiovasc Dev Dis. 2022 Oct 20;9(10):363. doi: 10.3390/jcdd9100363. PMID 36286314
- [Background] Akl E, Sahami N, Labos C, Genest J, Zgheib A, Piazza N, Jolly S. Meta-Analysis of Randomized Trials: Efficacy and Safety of Colchicine for Secondary Prevention of Cardiovascular Disease. J Interv Cardiol. 2024 Mar 12;2024:8646351. doi: 10.1155/2024/8646351. eCollection 2024. PMID 38505729
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Si HB, Yang TM, Zeng Y, Zhou ZK, Pei FX, Lu YR, Cheng JQ, Shen B. Correlations between inflammatory cytokines, muscle damage markers and acute postoperative pain following primary total knee arthroplasty. BMC Musculoskelet Disord. 2017 Jun 17;18(1):265. doi: 10.1186/s12891-017-1597-y. PMID 28623906
- [Background] Meert L, Mertens MG, Meeus M, Vervullens S, Baert I, Beckwee D, Verdonk P, Smeets RJEM. Identification of Metabolic Factors and Inflammatory Markers Predictive of Outcome after Total Knee Arthroplasty in Patients with Knee Osteoarthritis: A Systematic Review. Int J Environ Res Public Health. 2023 May 11;20(10):5796. doi: 10.3390/ijerph20105796. PMID 37239524
- [Background] Shah K, Mohammed A, Patil S, McFadyen A, Meek RM. Circulating cytokines after hip and knee arthroplasty: a preliminary study. Clin Orthop Relat Res. 2009 Apr;467(4):946-51. doi: 10.1007/s11999-008-0562-3. Epub 2008 Oct 22. PMID 18941856
- [Background] Zhang FS, He QZ, Qin CH, Little PJ, Weng JP, Xu SW. Therapeutic potential of colchicine in cardiovascular medicine: a pharmacological review. Acta Pharmacol Sin. 2022 Sep;43(9):2173-2190. doi: 10.1038/s41401-021-00835-w. Epub 2022 Jan 19. PMID 35046517
- [Background] Inturrisi CE. Clinical pharmacology of opioids for pain. Clin J Pain. 2002 Jul-Aug;18(4 Suppl):S3-13. doi: 10.1097/00002508-200207001-00002. PMID 12479250
- [Background] Chincholkar M. Analgesic mechanisms of gabapentinoids and effects in experimental pain models: a narrative review. Br J Anaesth. 2018 Jun;120(6):1315-1334. doi: 10.1016/j.bja.2018.02.066. Epub 2018 Apr 12. PMID 29793598
- [Background] Pepper AM, Mercuri JJ, Behery OA, Vigdorchik JM. Total Hip and Knee Arthroplasty Perioperative Pain Management: What Should Be in the Cocktail. JBJS Rev. 2018 Dec;6(12):e5. doi: 10.2106/JBJS.RVW.18.00023. No abstract available. PMID 30562208
- [Background] Kirwan MJ, Diltz ZR, Dixon DT, Rivera-Peraza CA, Gammage CJ, Mihalko WM, Harkess JW, Guyton JL, Crockarell JR, Ford MC. The AAHKS Clinical Research Award: Extended Postoperative Oral Tranexamic Acid in Total Knee Arthroplasty: A Randomized Controlled Pilot Study. J Arthroplasty. 2024 Sep;39(9S2):S13-S17. doi: 10.1016/j.arth.2024.02.073. Epub 2024 Feb 29. PMID 38430972
- [Background] Shaw JH, Wesemann LD, Banka TR, North WT, Charters MA, Davis JJ. The AAHKS Clinical Research Award: Oral Dexamethasone Following Total Knee Arthroplasty: A Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2023 Jul;38(7 Suppl 2):S15-S20. doi: 10.1016/j.arth.2023.04.046. Epub 2023 Apr 25. PMID 37105325
- [Background] Karam JA, Schwenk ES, Parvizi J. An Update on Multimodal Pain Management After Total Joint Arthroplasty. J Bone Joint Surg Am. 2021 Sep 1;103(17):1652-1662. doi: 10.2106/JBJS.19.01423. PMID 34232932
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Martinez GJ, Robertson S, Barraclough J, Xia Q, Mallat Z, Bursill C, Celermajer DS, Patel S. Colchicine Acutely Suppresses Local Cardiac Production of Inflammatory Cytokines in Patients With an Acute Coronary Syndrome. J Am Heart Assoc. 2015 Aug 24;4(8):e002128. doi: 10.1161/JAHA.115.002128. PMID 26304941
- [Background] Maniar RN, Navaneedhan G, Ranvir S, Maniar AR, Dhiman A, Agrawal A. What Is the Normal Trajectory of Interleukin-6 and C-reactive Protein in the Hours and Days Immediately After TKA? Clin Orthop Relat Res. 2019 Jan;477(1):41-46. doi: 10.1097/CORR.0000000000000332. PMID 30794227
- [Background] Kelly MP, Calkins TE, Culvern C, Kogan M, Della Valle CJ. Inpatient Versus Outpatient Hip and Knee Arthroplasty: Which Has Higher Patient Satisfaction? J Arthroplasty. 2018 Nov;33(11):3402-3406. doi: 10.1016/j.arth.2018.07.025. Epub 2018 Aug 1. PMID 30143333
- [Background] Hannon CP, Keating TC, Lange JK, Ricciardi BF, Waddell BS, Della Valle CJ. Anesthesia and Analgesia Practices in Total Joint Arthroplasty: A Survey of the American Association of Hip and Knee Surgeons Membership. J Arthroplasty. 2019 Dec;34(12):2872-2877.e2. doi: 10.1016/j.arth.2019.06.055. Epub 2019 Jul 8. PMID 31371038
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] Schwartz AM, Farley KX, Guild GN, Bradbury TL Jr. Projections and Epidemiology of Revision Hip and Knee Arthroplasty in the United States to 2030. J Arthroplasty. 2020 Jun;35(6S):S79-S85. doi: 10.1016/j.arth.2020.02.030. Epub 2020 Feb 19. PMID 32151524